CLINICAL TRIAL: NCT01740466
Title: Epidemiological Profile of Ophthalmological Care in the Public Service in Brazil
Acronym: EPP
Status: Completed | Type: Observational
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Other Study IDs: Epidemiological public profile
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Eye Abnormalities
Keywords: Prevalence; Vision disorders; Eye diseases; Visual acuity; Primary health care
MeSH Terms: conditions — Eye Abnormalities; Vision Disorders; Eye Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ocular diseases: Observational

SUMMARY:
Epidemiological study about eye discomfort complaints, comorbidities and diagnosis at a Brazil's ophthalmological public care service

DETAILED DESCRIPTION:
1. 1670 individuals underwent an ophthalmologic evaluation
2. The data were obtained through the analysis of the medical records with the ICD-10 registration
3. The studied variables were age and sex of patient, origin, eye discomfort complaints, comorbidities and diagnosis (ICD-10).
4. The purpose was to evaluate epidemiological aspects of eye diseases in a public service

ELIGIBILITY:
Inclusion Criteria:

* Patients assisted in public service

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals underwent an ophthalmologic evaluation
Sampling Method: Non-Probability Sample
Enrollment: 1670 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Incidence and prevalence of visual conditions in the Public Service in Brazil | 6 months
  * The ages ranged from 0 to 99 years
  * The mean age was 56.9 years
  * There was a predominance of females (58.1%)
  * The main reason for the consultation was low visual acuity (70%), followed by burning (26%) and itchiness (24.4%)
  * Among the abnormal tests there was a high prevalence of refractive errors (73.4%) and presbyopia (59.6%)
  * The cause of refractive errors was astigmatism (70.5%), hypertrophy (58.6%) and myopia (15.1%)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa N Figueiredo, Study Chair — IOG
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil